CLINICAL TRIAL: NCT04505046
Title: Validation of INSPiRED Innovative Smart Diagnostic Devices for the Detection of Plasmodium Falciparum, Schistosoma Haematobium and Necator Americanus at CERMEL, Gabon.
Brief Title: Validation of INSPiRED Innovative Smart Diagnostic Devices for the Detection of Parasites Infections.
Acronym: INSPiRED-WP3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CEI-005/2020
Record Dates: First submitted 2020-07-13; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Testing; Performance; Specificity; Sensitivity
Keywords: Plasmodium; Schistosoma; hookworm
MeSH Terms: conditions — Hypersensitivity; Malaria; Schistosomiasis; Ancylostomiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malaria, schistosomiasis and ancylostomiasis are three parasitic diseases which affect hundreds of millions of people and are an important cause of global mortality and morbidity. For the control of these poverty related parasitic diseases, and to complement chemotherapeutic strategies, accurate and accessible diagnostic procedures play a crucial role.

In recent years, innovative smart mobile technologies have been applied for detection and identification of cultured parasite species, which is basically based on sample imaging and parasite morphology identification. Promising advances have been made with this technology and coupled with its small size, low cost and easy to manipulate, makes it suitable for point of care diagnostics in low resource setting.

The aim of the proposed explorative study is to further validate sensitivity and specificity of each of the developed devices, using besides microscopy a range of more advanced reference tests.

DETAILED DESCRIPTION:
Malaria, schistosomiasis and ancylostomiasis are three parasitic diseases which affect hundreds of millions of people and are an important cause of global mortality and morbidity. For the control of these poverty related parasitic diseases, and to complement chemotherapeutic strategies, accurate and accessible diagnostic procedures play a crucial role. Especially in remote and/or low resource settings, appropriate diagnostic tests are often lacking. These tests should not only be sensitive and specific, but also affordable, reliable, and easy to operate. In recent years, innovative smart mobile technologies have been applied for detection and identification of cultured parasite species, which is basically based on sample imaging and parasite morphology identification. Promising advances have been made with this technology and coupled with its small size, low cost and easy to manipulate, makes it suitable for point of care diagnostics in low resource setting. At the Technical University of Delft, a smart optical device prototype has been recently developed for the detection of Plasmodium. This Excelscope has been tested on a small number of malaria cases in Nigeria, showing promising results. In addition, TU Delft has developed a prototype for the detection of Schistosoma haematobium eggs in urine, which is ready for further validation in the field. Still under construction is a smart optical device for the detection of helminth eggs in stool, including eggs of hookworms. For each of these three smart optical devices using respectively blood, urine or stool, a diagnostic performance is aimed which does not significantly deviate in sensitivity and specificity from the diagnostic tests commonly in use in low resource settings, e.g. basic microscopy. At the same time, the optical devices have supplementary logistical advantages, e.g. easiness to use, high throughput and low costs per sample. The aim of the proposed explorative study is to further validate sensitivity and specificity of each of the developed devices, using besides microscopy a range of more advanced reference tests. For this purpose, diagnostic samples (blood, urine, stool) collected from ongoing studies involving malaria, schistosomiasis and STHs. at CERMEL will be used. The outcome of this study will give new insight in the diagnostic performance of the innovative smart optical devices, specifically in comparison to the WHO recommended diagnostic procedures currently used at CERMEL. The study is the core activity of Work Package 3 within the INSPiRED project.

ELIGIBILITY:
Inclusion Criteria:

* Infected with malaria
* Infected with Schistosomiasis
* Soil-transmitted helminths

Exclusion Criteria:

-No sample provided

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All study participants, living in Lambaréné areas and its surrounding with parasitic infection
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
AiDx devise is good as a conventional microscopy | 3 years
  Optical diagnostic devices is specific, sensitive as well as predicting value as microscopic test
Schistoscope | 3 years
  Optical diagnostic devices is specific, sensitive as well as predicting value as microscopic test
Hookworm and other STH devise is good as conventional. microscopic test | 3 years
  Optical diagnostic devices is specific, sensitive as well as predicting value as microscopic test

CONTACTS AND LOCATIONS:
Overall Officials: Romuald Mba, MSc, Study Chair — Centre de Recherches Médicales de Lambaréné - CERMEL
Locations (1):
- Centre de Recherches Medicales de Lambarene, Lambaréné, Moyen-Ogooué Province, Gabon

REFERENCES:
- [Derived] Meulah B, Oyibo P, Hoekstra PT, Moure PAN, Maloum MN, Laclong-Lontchi RA, Honkpehedji YJ, Bengtson M, Hokke C, Corstjens PLAM, Agbana T, Diehl JC, Adegnika AA, van Lieshout L. Validation of artificial intelligence-based digital microscopy for automated detection of Schistosoma haematobium eggs in urine in Gabon. PLoS Negl Trop Dis. 2024 Feb 23;18(2):e0011967. doi: 10.1371/journal.pntd.0011967. eCollection 2024 Feb. PMID 38394298